CLINICAL TRIAL: NCT04516083
Title: Correlation Between Somatic Mismatch Repair Instability and Germline Mismatch Repair Instability, in Low Socioeconomic Background Population Diagnosed With Endometrial Endometrioid Adenocarcinoma
Brief Title: Lynch Syndrome Can be Diagnosed Just From Somatic Mismatch Repair Mutation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: RWJ Barnabas Health at Jersey City Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 1272883
Record Dates: First submitted 2020-08-03; First posted 2020-08-17 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Cancer Gene Mutation; Lynch Syndrome; Endometrial Cancer; Somatic Mutation
MeSH Terms: conditions — Colorectal Neoplasms, Hereditary Nonpolyposis; Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Mismatch repair instability somatic and germline testing — Each Endometrial Endometrioid adenocarcinoma is routinely stained for MMR mutation to seek for tumor genetic instability. If stains positive, the patient is called in for genetic blood testing to look for the same mutation in the germline.

SUMMARY:
The objective of the study is the provide proof of high correlation between somatic and germline mismatch repair instability. This correlation is specifically researched in an area where patients have less access to cancer education and genetic testing for various reasons such as lack of insurance and general accessibility.

The study concentrates on early diagnosis of Lynch syndrome. Lynch syndrome is usually diagnosed from a blood test resulting in a mutation of one of the mismatch repair genes. Those are MLH1, MSH2, MSH 6, PMS2. A mutation in one of these genes creates a mismatch repair instability,hence higher incidence of cancers in specific organ groups. Amongst these organs are the Uterus, Ovaries, Upper genitourinary system, Pancreas and GI system.

The most common endometrial carcinoma which is found in Lynch syndrome is of endometrioid histology. Most patients with known germline mismatch repair instability, have the same somatic mutation. Our study is looking into correlating somatic mutation to germline mutation.

By doing so, patients diagnosed with somatic mismatch repair instability will be also diagnosed with lynch syndrome without germline genetic testing.

Screening programs will be utilized earlier and preventive procedures offered.

Due to less access to educational programs, genetic counseling and testing in underserved areas, patients are sometimes lost to follow up. Our study seeks to prove high correlation between somatic and germline mutations and by doing so, patient will be diagnosed with Lynch syndrome straight after endometrial cancer staging. As a result, increased compliance will be expected and patients will be offered the recommended preventative surgeries and screening protocols.

ELIGIBILITY:
Inclusion Criteria:

Underserved areas. Diagnosis of endometrial endometrioid carcinoma. Low socioeconomic status. Positive mismatch repair staining. All races. All ages. All cancer grades. All cancer stages .

Exclusion Criteria:

Diagnosis of type 2 endometrial carcinoma. Cancer diagnosis other than Endometrial. No mismatch repair genes mutation. High socioeconomic status.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Female as this is endometrial carcinoma
Study Population: The population includes female patients of all ages and races who are from a low socioeconomic background defined by the american psychological association.
  These females usually reside in underserved area. All the patients are diagnosed with endometrial endometrioid adenocarcinoma via tissue biopsy.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-12-21 (Actual); Primary Completion 2020-12-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of patients who have a somatic mutation at the same time as a germline mutation | Through study completion, an average of 18 months
  1. Resected tissue during endometrial staging will be immunohistochemically stained for MMR mutation.
  2. Patient blood test will be checked for MMR gene mutation
  3. Linear regression curve will be constructed to evaluate the correlation between somatic and germline mutation.

CONTACTS AND LOCATIONS:
Locations (1):
- Jersey city medical center, Jersey City, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chu MM, Liu SS, Tam KF, Ip PP, Cheung AN, Ngan HY. The Significance of Mismatch Repair Deficiency in Young Patients With Endometrial Cancer. Int J Gynecol Pathol. 2015 Sep;34(5):403-10. doi: 10.1097/PGP.0000000000000174. PMID 26262451
- [Background] Modica I, Soslow RA, Black D, Tornos C, Kauff N, Shia J. Utility of immunohistochemistry in predicting microsatellite instability in endometrial carcinoma. Am J Surg Pathol. 2007 May;31(5):744-51. doi: 10.1097/01.pas.0000213428.61374.06. PMID 17460459
- [Background] Kahn RM, Gordhandas S, Maddy BP, Baltich Nelson B, Askin G, Christos PJ, Caputo TA, Chapman-Davis E, Holcomb K, Frey MK. Universal endometrial cancer tumor typing: How much has immunohistochemistry, microsatellite instability, and MLH1 methylation improved the diagnosis of Lynch syndrome across the population? Cancer. 2019 Sep 15;125(18):3172-3183. doi: 10.1002/cncr.32203. Epub 2019 May 31. PMID 31150123